CLINICAL TRIAL: NCT05601336
Title: Effect of Sodium Glucose Cotransporter-2 Inhibitors on Metabolic, Hormonal and Clinical Parameters in Infertile Women With Polycystic Ovary Syndrome
Brief Title: of Sodium Glucose Cotransporter-2 Inhibitors on Metabolic, Hormonal and Clinical Parameters in PCO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-22012
Record Dates: First submitted 2022-10-15; First posted 2022-11-01 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: PCO
MeSH Terms: interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- metformin monotherapy (Active Comparator): Glucophage 1000 once daily
  Interventions: Drug: Metformin Hydrochloride 1000 MG
- Dapagliflozin monotherapy . (Active Comparator): Farxiga once per day
  Interventions: Drug: Dapagliflozin 5 MG
- metformin and dapagliflozin combined therapy (Active Comparator): Xigduo once daily
  Interventions: Drug: Dapagliflozin/Metformin
- control group. (No Intervention): placebo

INTERVENTIONS:
Drug: Dapagliflozin 5 MG — SGLT2 inhibitor
  Other Names: [Farxiga]
  Arms: Dapagliflozin monotherapy .
Drug: Metformin Hydrochloride 1000 MG — metformin
  Other Names: Glucophage 1000mg
  Arms: metformin monotherapy
Drug: Dapagliflozin/Metformin — SGLT2 inhibitor and metformin HCl extended-release
  Other Names: Xigduo
  Arms: metformin and dapagliflozin combined therapy

SUMMARY:
The aim of this study is to compare the hormonal, metabolic and clinical effects of metformin and dapagliflozin as monotherapies and the effect of both of them as a combined therapy in infertile women with PCOs.

DETAILED DESCRIPTION:
It is a Prospective randomized controlled trial .The study will include 200 randomly selected infertile women aged between 18 and 45 years, from Gynecology and obstetrics department Beni-Suef University Hospital whom diagnosed with polycystic ovarian syndrome (PCOS), according to Rotterdam criteria (BMI≥ 24kg/m, Homeostatic model assessment of insulin resistance (HOMA-IR with cutoff ≥ 2.5 biochemical hyperandrogenism, as indicated by a free androgen index (FAI) >4, and self-reported oligomenorrhea (cycle length >35 days and 9 or fewer periods per year) or amenorrhoea (absence of menses for a period ≥3 months) will be included for the study.

I The study will include four groups; each group consists of 50 patients:-

* Group I (n=50) will be treated by metformin monotherapy.
* Group II (n=50) will be treated by Dapagliflozin monotherapy .
* Group III (n=50) will be treated by metformin and dapagliflozin combined therapy
* Group IV (n=50) will be a control group.

ELIGIBILITY:
Inclusion Criteria:

* Women are aged between 18 and 45 years
* no pregnancy plan within the next 6 months
* polycystic ovarian syndrome (PCOS), according to Rotterdam criteria

Exclusion Criteria:

1. congenital adrenal hyperplasia
2. poorly controlled thyroid disease
3. Taking antidiabetic drugs which can affect insulin resistance
4. chronic kidney disease and history of recurrent urinary tract infections
5. liver dysfunction (AST or ALT > 3 times the upper limit of normal or GFR<30 ml/min/1.73m2)
6. documented use of oral hormonal contraceptives and hormone-releasing implants

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
ovulation | 3 cycles ( 3 months / one month for each cycle)
  folliculometry by ultrasound
Cummulative rate of pregnancy | 3 months
  HCG test

SECONDARY OUTCOMES:
Body weight changes | 3 months
  weight loss by Kg
changes of Menstrual cycle | 3 months
  history from the patient
Fasting blood sugar (FBS)/ 2 hpp | 3 months
Free Androgen Index (FAI) | 3 months
Total Testosterone (TT) | 3 months
FSH*LH*E2 | 3 months
lipid profile | 3 months
ALT | 3 months
side effects | 3 months
  Number of patients will report nausea / diarrhea/ lactic acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Study Director — Clinical Pharmacy Faculty of Pharmacy Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: within 36 months